CLINICAL TRIAL: NCT03078283
Title: Effects of High-fiber Snack Foods on Human Gut Microbes
Brief Title: Food Effects on the Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Mondelēz International, Inc. (Industry)
Responsible Party: Principal Investigator, Jeffrey I. Gordon, Dr. Robert J. Glaser Distinguished University Professor, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MDLZ2017JIG1
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Gut Microbial Responses to Dietary Fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Consumption of a given type of high-fiber snack food, with each individual functioning as her own control
  Interventions: Other: high-fiber food type

INTERVENTIONS:
Other: high-fiber food type — In 3 successive experiments, usual diet will be supplemented with snack foods containing fiber of plant, fruit or grain origin.

SUMMARY:
This is a small-scale study of the effects on microbes in the human gut of adding high-fiber snack foods to usual diet. The snack foods are being provided by Mondelez International, Inc. Eight pairs of dizygotic twins, discordant or concordant for obesity, will participate in the study. They will complete 3 successive experiments in which their regular diet is supplemented by consumption, over a 6-week period, of high-fiber snack foods. Each experiment will involve (i) two weeks consuming regular diet (fecal sample collected weekly); (ii) one week consuming one snack food per day (approximately 7 g fiber, collection of all fecal samples), (iii) one week consuming two snack foods per day (approximately 14 g fiber, collection of all fecal samples), (iv) four weeks consuming three snack foods per day (approximately 20 g fiber, collection of all fecal samples); and (v) two weeks consuming only regular diet (weekly collection of fecal sample). For each experiment, participants will also provide a fasting blood sample during the free diet phase at the end of the week just before initiation of snack consumption, and a fasting blood sample at the end of the last week of snack consumption. Participants will also collect one first morning urine sample weekly throughout the study. During week 2, participants will also collect first morning urine samples for 3 consecutive days. Similarly, they will collect first morning urine samples for the last 3 consecutive days of the last week of snack consumption. The study will test the effects of the different fiber-rich snacks on the composition and metabolic properties of the gut microbial community in lean and obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* member of female dizygotic twin pair discordant or concordant for obesity

Exclusion Criteria:

* pregnant or trying to get pregnant
* inflammatory bowel disease
* gastrointestinal cancer
* hepatitis
* HIV
* renal failure
* food allergies

Ages: 31 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Assessment of gut microbial community structure and function | 8 weeks
  Sequencing bacterial 16S rRNA amplicons plus shotgun sequencing of fecal community DNA to identify effects of fiber-enriched foods on bacterial community and gene representation; mass spectrometry of products of gut microbial community metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Gordon, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual data will be shared after completion of the study, to the extent that this can be accomplished without violating the confidentiality of participants (some of whom would be easily identifiable from their clinical metadata).

REFERENCES:
- [Background] Ridaura VK, Faith JJ, Rey FE, Cheng J, Duncan AE, Kau AL, Griffin NW, Lombard V, Henrissat B, Bain JR, Muehlbauer MJ, Ilkayeva O, Semenkovich CF, Funai K, Hayashi DK, Lyle BJ, Martini MC, Ursell LK, Clemente JC, Van Treuren W, Walters WA, Knight R, Newgard CB, Heath AC, Gordon JI. Gut microbiota from twins discordant for obesity modulate metabolism in mice. Science. 2013 Sep 6;341(6150):1241214. doi: 10.1126/science.1241214. PMID 24009397